# STATISTICAL ANALYSIS PLAN (SAP)

# **Project Title**

A multicenter, single blind, randomized controlled trial of virucidal effect of Polyvinylpyrrolidone-Iodine on SARS-CoV-2 as well as safety of its application on nasopharynx & oropharynx of COVID-19 positive patients

BMRC Reg. No: 38624012021

## **Statistical Analysis Plan (SAP)**

## 1. Sampling Technique

Sample Size

• The minimum sample size is given by:

Where, n= sample size Z= Standard normal deviate usually set at 1.96 at 95% confidence If prevalence is not known, the value of prevalence will be considered as 50%.

So, p will be 0.5.

So, 
$$q = (1-p) = 0.50$$
, and

d = Desired accuracy or degree of allowable error. It is usually set as 5%(0.05).

So, 
$$n = \{(1.96)2 \times 0.5 \times 0.5\} / (0.05)2$$

Or, 
$$n = 384$$

for a finite population  $n = (Z2 \times p \times q) / d2$ 

N.B. Calculated sample size is equally applicable for both experimental (Intervention) and control group.

## 2. Statistical Analysis tools

Data analysis software : Statistical Package for the Social Sciences (SPSS)

Descriptive statistical parameter : Mean, Medium, Mode, Standard Deviation, Percentage,

Frequency

Inferential statistics : Chi-square test, t-tes, F-test, Anova, Correlation

Confidence Interval : 95%